CLINICAL TRIAL: NCT04625023
Title: A Master Protocol Empowering Mechanobiology Translation Research in Breast Cancer
Acronym: METAMECH
Status: Recruiting | Type: Observational
Sponsor: IFOM ETS - The AIRC Institute of Molecular Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IFOM-CPO007/2019/PO006
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — * FFPE tissue
  * Fresh Tissue (tumor and normal)
  * Plasma
  * PBMC
  * Whole Blood
  * Stools
  * Buccal Swabs
  * Pleural effusions and ascites
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort of BC patients: Stage-mixed cohort of at least 1500 breast cancer patients through their course of treatment, until death or a minimum of 5 years.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Retrospective cohorts and Prospective observation of standard clinical practice

SUMMARY:
METAMECH is a master observational protocol designed to empower a bi-directional collaboration between basic and clinical research, an essential prerequisite to feed and implement precision oncology.

METAMECH will follow a stage-mixed cohort of at least 500 patients through their course of treatments, until death or a minimum of 5 years. Patients will be longitudinally sampled and matched clinical data (including imaging) will be collected. Via a multi-tiered informed consensus process, METAMECH will also allow to develop companion diagnostics for molecular enrichment strategies in AIRC-driven proof-of-concept trials.

DETAILED DESCRIPTION:
METAMECH has been designed to streamline the study of the co-evolutionary landscape between tumor and host cells in a cohort of breast cancer (BC) patients, with the aim of understanding how their outcomes can be significantly improved (e.g. reduction of their chance of recurrence and survival improve). This clinical resource for integrative clinical data and sample collection will allow to generate hypotheses on mechanisms supporting the outgrowth of human metastases, mine for new potentially actionable targets and the selection of appropriate patients for experimentally-driven trials. To achieve the required level of 'experimental precision', patients will enter METAMECH at two different 'therapeutic checkpoints': i) prior to a tumor sampling event (surgery, biopsy) or ii) prior to any line of treatment.

To optimize the enrollment of patients, the longitudinal collection of data/samples and their logistic management, METAMECH has been designed as a flexible infrastructure organized in Tiers for the stepwise comprehension of the biological processes that drive tumor evolution, and precisely:

* TIER0, Retrieving: the ability to retrospectively retrieve clinically annotated BC archival samples to validate/discover new mechanotransduction-linked biomarkers;
* TIER1, Recording: the ability to prospectively record BC characteristics under standard of care treatments and to define new mechanotransduction-linked biomarkers;
* TIER2, Modelling: the ability to develop pertinent experimental models to study the aberrant mechanisms underlying the metastatic outgrowth and define mechanotransduction-targeting therapeutic strategies;
* TIER3, Linking: the ability to access data and samples of patients enrolled in POC trials to prove the efficacy and study/understand resistance mechanisms of mechanotransduction-targeting therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Verification that the patient could not be reached for informed consent in accordance with applicable national regulations or, alternatively, TIER1 written Informed consent.
2. Patients ≥18 years of age.
3. Previous diagnosis of breast cancer, or a strong suspicion of BC based on clinical and radiological findings.
4. ECOG Performance status < 2 (only for TIER1-2).

Exclusion Criteria:

1. Any other current malignancy or malignancy diagnosed or relapsed within the past 5 years (other than non-melanomatous skin cancer, stage 0 melanoma in situ, and in situ cervical cancer)
2. Patient unable to comply with the study protocol owing to psychological, social or geographical reasons.
3. Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) or syphilis infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage-mixed Breast Cancer (BC) patients
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-07-16 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients recruited in TIER0 and TIER 1 | 6 months
  Number of recruited BC cases in TIER 0 and in TIER 1 with complete clinically annotated FFPE and/or frozen biological samples
Number of patients recruited in TIER2 | 6 months
  Number of recruited BC cases in TIER 2

SECONDARY OUTCOMES:
Number of patients triaged in proof-of concept (POC) clinical trials | 6 months
  Number of BC cases recruited in TIER 3

OTHER OUTCOMES:
New prognostic mechanotransduction-linked markers | 6 months
  Number of identified/validated new prognostic mechanotransduction-linked markers
New predictive mechanotransduction-linked markers | 6 months
  Number of identified/validated new predictive mechanotransduction-linked markers
Biomarkers correlation with RR | 6 months
  Correlation between identified biomarkers with therapies response rates (RR)
Biomarkers correlation with PFS | 6 months
  Correlation between identified biomarkers with progression-free survival (PFS)
Biomarkers correlation with OS | 6 months
  Correlation between identified biomarkers with overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Marsoni, MD, Study Chair — IFOM ETS - The AIRC Institute of Molecular Oncology
Locations (10):
- Italy (10):
  - Asst Papa Giovanni Xxiii, Bergamo, Bergamo
  - Fondazione IRCCS, Istituto Nazionale dei Tumori, Milan, Milan
  - Fondazione IRCCS, Istituto Neurologico Carlo Besta, Milan, Milan
  - Azienda Ospedaliero Universitaria Maggiore della Carità di Novara, Novara, Novara
  - Istituto Oncologico Veneto IRCCS (IOV), Padua, Padova
  - Fondazione IRCCS, Policlinico San Matteo Pavia, Pavia, Pavia
  - Istituto Nazionale Tumori Regina Elena di Roma - Istituti Fisioterapici Ospitalieri (IFO), Roma, Roma
  - IRCCS Humanitas, Milan
  - IEO - Istituto Europeo di Oncologia, Milan
  - Azienda U.S.L. - IRCCS di Reggio Emilia, Reggio Emilia

IPD SHARING:
Plan to Share IPD: Undecided